CLINICAL TRIAL: NCT00776932
Title: Disparity in Joint Replacement: Pathway to Intervention
Brief Title: Chronic Knee Pain Study
Acronym: JRPIT
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 07040263; 1 P60 AR05473-01
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Knee OA: Those over the age of 50 who have frequent pain in their knee that has lasted for at least six months.

SUMMARY:
Specific Aims: 1) To examine differences between AA and white patients with knee OA in willingness to consider knee joint replacement. 2) To examine the relationship between socio-cultural factors and patient willingness to consider joint replacement. 3) To examine how demographic, socio-cultural, and clinical factors mediate the relationship between race and patient willingness. 4) To examine the relationship between patient willingness and referral to orthopedic care for knee OA (secondary aim).

Experimental design/Methodology: A cross-sectional survey study design will be used to examine socio-cultural and clinical factors that may vary by race/ethnicity and may be determinants of willingness to consider joint replacement as a treatment option. Patients with symptomatic and radiographic knee OA from the primary care clinics will be surveyed. Only individuals with knee OA of sufficient severity that would be considered candidates for joint replacement will be included. Analytic strategies include ordinal logistic regression, path analysis, and regression trees.

Subject population: The study sample will consist of approximately 133 African American and 419 white patients with OA of the knee in a primary care setting.

ELIGIBILITY:
Inclusion Criteria:

* over age 50
* chronic knee pain
* radiographic evidence of knee OA

Exclusion Criteria:

* previous joint replacement
* inflammatory arthritis

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: African Americans and Whites over the age of 50 with chronic knee pain.
Sampling Method: Non-Probability Sample
Enrollment: 852 (Actual)
Dates: Start 2007-06; Primary Completion 2011-08 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Compared to whites, AAs with knee OA will be less willing to consider joint replacement. Logistic regression will be used to model the categorical measure of willingness, if preliminary analyses indicate dichotomizing this measure. | Study Completion

CONTACTS AND LOCATIONS:
Overall Officials: C. Kent Kwoh, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburh Arthritis Research Center, Pittsburgh, Pennsylvania, United States